CLINICAL TRIAL: NCT03048994
Title: A Randomized Controlled Trial of Glutamine Supplementation in Critically Ill Adults With Severe Sepsis: A Pilot Study
Brief Title: Glutamine Supplementation in Critically Ill Patients With Severe Sepsis
Acronym: CGH-GLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTC1000338
Record Dates: First submitted 2012-09-24; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Severe Sepsis
Keywords: Glutamine; Severe sepsis
MeSH Terms: conditions — Sepsis | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Glutamine (Active Comparator): Glutamine
  Interventions: Dietary Supplement: Glutamine

INTERVENTIONS:
Dietary Supplement: Glutamine — * Patients randomised to receive glutamine supplementation will receive IV glutamine (0.5g/kg body weight/day) continuously over 24 hours.
  * IV glutamine will be administered for 5 days or less if death ensues prior to 5 days or transferred to another hospital prior to 5 days. IV glutamine will be continued even if the patient is transferred outside the ICU but within the hospital.
  * An intravenous saline solution that is identical in volume, color and consistency will be administered to the placebo group with the same dosing regimen and duration.
  Arms: Glutamine
Dietary Supplement: Placebo — * Nutritional support will be continued as per managing ICU team discretion.
  * Management of severe sepsis will be continued as per managing ICU team discretion.
  * Weaning patients from mechanical ventilation will be done as per managing ICU team discretion.
  * To minimise differences between centers, active dissemination of practice guidelines for nutritional support, sepsis management and weaning will be carried out.
  Arms: Placebo

SUMMARY:
Severe sepsis is a common condition with high mortality and morbidity. A previous meta-analysis has demonstrated the safety of glutamine supplementation with suggestion of mortality and morbidity benefits in critically ill patients. But there is lack of evidence to recommend the use of intravenous glutamine supplementation in this population group. A randomized controlled trial which is adequately powered will resolve this issue and can be included in future international nutrition guidelines for the critically ill. This pilot study is done prior to a proposed local multi-center study to investigate the effects of glutamine supplementation.

DETAILED DESCRIPTION:
Objective

* To determine the effect of intravenous glutamine supplementation compared with placebo in critically ill patients with severe sepsis
* Primary outcome : 28 day mortality , Development of infectious complications
* Secondary outcomes

  * Duration of mechanical ventilation
  * Length of stay in ICU
  * Length of stay in hospital
  * 3 month survival status and resumption of baseline activities
  * 6 month survival status and resumption of baseline activities

Study Design

* Single center, prospective, double blind, randomised controlled trial critically ill patients with severe sepsis
* Randomisation

  * A centralised randomisation system at SCRI (Singapore Clinical Research institute)
  * Allocation will be random and concealed, and will be blinded to everyone except the pharmacist at each site, who will be responsible for preparing and delivering them to the ICU in a blinded fashion.
* Intervention

  * Patients randomised to receive glutamine supplementation will receive IV glutamine (0.5g/kg body weight/day) continuously over 24 hours.
  * IV glutamine will be administered for 5 days or less if death ensues prior to 5 days or transferred to another hospital prior to 5 days. IV glutamine will be continued even if the patient is transferred outside the ICU but within the hospital.
  * An intravenous saline solution that is identical in volume, color and consistency will be administered to the placebo group with the same dosing regimen and duration.
* Cointerventions

  * Nutritional support will be continued as per managing ICU team discretion.
  * Management of severe sepsis will be continued as per managing ICU team discretion.
  * Weaning patients from mechanical ventilation will be done as per managing ICU team discretion.
  * To minimise differences between centers, active dissemination of practice guidelines for nutritional support, sepsis management and weaning will be carried out.

Execution of study protocol

* The managing ICU team will be responsible in identifying patients that meet the inclusion and exclusion criteria and will inform the site research coordination
* The site research coordinator will be responsible for the following

  * Obtaining consent from relatives of the patients
  * Informing the site pharmacist about the recruited patients
  * Follow study patients prospectively while in the ICU, hospital and post discharge at 3 and 6 months.
  * Completing the case report from for each study participant
  * Submitting case report forms, completed and interim reports, to coordinating statistical team
* Pharmacist

  * Site pharmacist to liase with SCRI on randomised patients status (treatment vs. placebo)
  * Prepare the intervention treatment and placebo
  * Deliver the treatment and placebo to the respective patients.
* Nurses

  * Responsible for administering the delivered medications
  * Ensure and documenting compliance with administration, reasons for interruptions and documenting adverse reactions.
  * Liasing with the site research coordinator daily regarding the above.
  * Liasing with the site research coordinator on transfer, discharge or death of study participants

ELIGIBILITY:
Inclusion Criteria

* All adult patients (>18 years old) admitted to ICU plus
* Severe sepsis defined as 2 or more or the following

  * Temperature >38oC or < 36oC
  * Heart rate > 90 beats per min
  * Respiratory rate >20 breaths per min or PaCO2 <32 mmHg
  * White cell count > 12,000/microL or < 4,000/microL

    * PLUS presence or presumed presence of infection
    * PLUS evidence of organ dysfunction as defined by either of the following
    * Hemodynamic: Hypotension = systolic blood pressure (SBP) 40 mm Hg or mean arterial pressure (MAP) < 65 mm Hg; or on vasopressors
    * Hyperlactatemia: Serum lactate >/= 2 mmol/L (18 mg/dL)
    * Renal: Acute increase in serum creatinine to > 176.8 mmol/L (2.0 mg/dL) or urine output < 0.5 mL/kg/hour for > 2 hours
    * Lung: Acute lung injury with PaO2/FiO2 </=300mmHg
    * Liver: Acute increase in bilirubin to >/= 34.2 umol/L (2 mg/dL)
    * Thrombocytopenia: Acute decrease in platelet count to < 100,000 cells/mm3
    * Coagulopathy: International normalized ratio (INR) > 1.5 or a partial thromboplastin time (aPTT) > 60 secs which is not due to anticoagulant therapy
  * Exclusion criteria
* >48hr from admission to ICU
* Patients who are not expected to survive >48hrs by the managing team
* Refusal to consent to study
* Allergic to glutamine or its constituents
* Absolute contraindication to enteral nutrition or the need to initiate parenteral nutrition
* Patients with a primary admission diagnosis of burns (>30% body surface area)
* Patients whose weight <40kg or >200kg
* Previous randomization to this study
* Enrolled in a related ICU interventional nutrition study
* Pregnant patients or lactating mothers with the intent to breastfeed

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 day

SECONDARY OUTCOMES:
Occurrence of new infections | Initial hospital admission, assessed up to 130 days.
ICU length of stay (LOS) | From date of ICU admission to date of transferred to General Ward or date of death from any cause, whichever came first, assessed up to 21 days.
Hospital LOS | From date of recruitment to date of discharged from hospital or date of transferred to other hospitals or date of death from any cause, whichever came first, assessed up to 130 days.
Duration of mechanical ventilation | During period of ICU stay, assessed up to 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Vijo Poulose, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novak F, Heyland DK, Avenell A, Drover JW, Su X. Glutamine supplementation in serious illness: a systematic review of the evidence. Crit Care Med. 2002 Sep;30(9):2022-9. doi: 10.1097/00003246-200209000-00011. PMID 12352035
- [Background] Roth E, Funovics J, Muhlbacher F, Schemper M, Mauritz W, Sporn P, Fritsch A. Metabolic disorders in severe abdominal sepsis: glutamine deficiency in skeletal muscle. Clin Nutr. 1982 Mar;1(1):25-41. doi: 10.1016/0261-5614(82)90004-8. PMID 16829366
- [Background] Heyland DK, Dhaliwal R, Suchner U, Berger MM. Antioxidant nutrients: a systematic review of trace elements and vitamins in the critically ill patient. Intensive Care Med. 2005 Mar;31(3):327-37. doi: 10.1007/s00134-004-2522-z. Epub 2004 Dec 17. PMID 15605227